CLINICAL TRIAL: NCT04587947
Title: Influence of Sacubitril/Valsartan on Autonomic Cardiac Nervous System in Heart Failure Patients: an Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Entresto
Record Dates: First submitted 2020-06-24; First posted 2020-10-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure Patients
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Heart rate variability measurement is carried out by means of a 12-channel ECG for 30 minutes in supine position followed by 10 minutes in standing position. All parameters, including blood values and echocardiographic parameters are assessed before beginning of sacubitril/ valsartan therapy and 3 months after starting treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sacubitril/ valsartan — Heart rate variability measurement is carried out by means of a 12-channel ECG for 30 minutes in supine position followed by 10 minutes in standing position. All parameters, including blood values and echocardiographic parameters are assessed before beginning of sacubitril/ valsartan therapy and 3 months after starting treatment

SUMMARY:
Sacubitril/valsartan is an angiotensin receptor neprilysin inhibitor with the ability to reduce myocardial hypertrophy, cardiac remodeling and cardiorenal fibrosis. The compound is also believed to have antiarrhythmic properties as it has been shown to significantly reduce ventricular arrhythmias in patients with implantable cardioverter defibrillators.

Patients suffering from heart failure with reduced ejection fraction show impaired heart rate variability, knowing that in these patients such impairment is highly associated with an increased risk of sudden cardiac death.

In its pivotal study, sacubitril/valsartan demonstrated a significant advantage over enalapril in terms of cardiovascular mortality and rehospitalization.

Against this background, this study was designed to analyze the largely unknown electrophysiological effects of sacubitril/valsartan on the autonomic cardiac nervous system by determining heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic severe heart failure with reduced ejection fraction (LVEF ≤40%,)
* Age > 20 years
* Consent capacity
* Sinus rhythm
* Suitable for a drug conversion from AT1/ACE inhibitors to sacubitril/ valsartan

Exclusion Criteria:

* Age < 18 years
* Atrial fibrillation
* Pregnancy
* Lack of consent capacity
* Contraindications for a therapy with sacubitril/ valsartan

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability | 24 months
  Changes in heart rate variability after 3 months of treatment with sacubitril/ valsartan
Changes in left ventricular ejection fraction (%) | 24 months
  Changes in left ventricular ejection fraction (%) assessed by transthoracic echocardiogramChanges in echocardiographic parameters (left ventricular parameters)
Changes in mitral insufficiency grade | 24 months
  Changes in mitral insufficiency grade assessed by transthoracic echocardiogram
Changes in serum NT-proB-Type natriuretic peptide (ng/l) | 24 months
  Changes in laboratory parameters (serum NT-proB-Type natriuretic peptide (ng/l)
Changes in Serum creatinine level (mg/dl) | 24 months
  Changes in laboratory parameters (Serum creatinine level (mg/dl)
Changes in glomerular filtration rate (ml/min) | 24 months
  Changes in laboratory parameters (glomerular filtration rate ml/min)
Changes in serum potassium level (mmol/l) | 24 months
  Changes in laboratory parameters (glomerular filtration rate ml/min)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden, Germany

REFERENCES:
- [Result] Boehmer AA, Schubert T, Rothe M, Keim C, Wiedenmann L, Ruckes C, von Stuelpnagel L, Theurl F, Schreinlechner M, Dobre BC, Kaess BM, Bauer A, Ehrlich JR. Angiotensin Receptor-Neprilysin Inhibitor Is Associated With Improved Cardiac Autonomic Function in Heart Failure. J Am Heart Assoc. 2024 Aug 6;13(15):e033538. doi: 10.1161/JAHA.123.033538. Epub 2024 Jul 31. PMID 39082399